CLINICAL TRIAL: NCT01407419
Title: Treating to Target (T2T) for Patients With Rheumatoid Arthritis in a US Population: Outcomes and Feasibility
Brief Title: The CORRONA Treat to Target Trial: Outcomes and Feasibility in a US Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEIRB 11-216
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treat to Target Intervention Strategy (Experimental): Subjects at sites randomized to this arm will be expected to return to the clinic for Monthly Assessments until low disease activity (LDA) defined as CDAI of 10 or less has been achieved. Providers are prompted to accelerate therapy (Treatment Acceleration) at each visit that CDAI is >10 (unless not felt to be medically appropriate or refused by the subject.) Accelerations are expected at least every 3 months, until/unless LDA has been achieved.
  Interventions: Other: Treatment Acceleration; Other: Monthly Assessment
- Control Group Treated with Usual Care (No Intervention): Subjects in this arm will be expected to complete study visits with their rheumatologist/study doctor at Baseline, Month 3, Month 6, Month 9 and Month 12. Data collection will occur at each of those visits. Subjects and Providers will continue managing disease per usual practices and do not receive protocol prompts relative to visit frequency or acceleration of therapy, regardless of disease activity level (by CDAI)

INTERVENTIONS:
Other: Treatment Acceleration — Subjects in the intervention group will be seen as frequently as monthly for subjects not achieving low disease activity (LDA) as defined as CDAI ≤10. Treatment acceleration will be expected to occur as frequently as monthly and at least every 3 months in these subjects, unless contraindicated.
  Treatment acceleration for the purposes of this trial include the following options: Change in prescribed treatment or dosage of "traditional" or "biologic" Disease Modifying Anti Rheumatic Drugs (DMARDs) or a change in the route of Methotrexate administration (from oral to subcutaneous)
  Arms: Treat to Target Intervention Strategy
Other: Monthly Assessment — Monthly disease assessments are expected to be scheduled until the subject has achieved a CDAI of 10 or less (low disease activity).
  Other Names: Monthly follow-up visits to rheumatologist
  Arms: Treat to Target Intervention Strategy

SUMMARY:
The Treat to Target Trial is a clinical trial available to new and existing CORRONA (Data Collection Program) sites. Subjects are recruited to participate in this 12 month trial examining outcomes and feasibility of implementing a Treat to Target approach, when compared with a control group of subjects treated with usual care.

DETAILED DESCRIPTION:
New and existing CORRONA sites and patient participants are recruited to participate as subjects in this 12 month trial examining outcomes and feasibility of implementing a Treat to Target approach to RA disease management, requiring routine monthly monitoring and regular escalations of treatment for subjects not achieving low disease activity (LDA) when compared with a control group of subjects treated with usual care.

Purpose The primary purpose of the study is to determine whether practices implementing a multi-dimensional T2T process can more effectively control active Rheumatoid Arthritis (RA) in patients eligible-for-acceleration compared to those practices which continue usual care. The trial will also determine if the process of treating to target for the selected subjects is different between the two groups.

A wide variety of therapies are used in clinical practice to treat patients with RA. The CORRONA Data Collection Program is designed to collect and document utilization patterns, effectiveness, and safety of DMARDs (Disease Modifying Anti-Rheumatic Drugs), biologic agents, and many other treatments currently used in the management of rheumatic diseases. It is anticipated that the study data may help improve the quality of information upon which clinical decisions are based.

Objectives Co-primary Objectives 1. To measure rates of low disease activity (by CDAI score) between treatment arms (T2T vs usual care) at 12 months.

1a. To assess implementation of a T2T Protocol by comparing rates of acceleration, frequency of visits, time to next visit, and probability of acceleration conditional on disease activity between subjects treated in a T2T intervention group, compared with a control group treated with usual care (UC) at 12 months.

Secondary Objectives

1. To determine mediators of differences in LDA rates between the two randomized groups.
2. To determine the association between the process of treating to target and LDA (regardless of randomization).
3. To determine the proportion of subjects with active RA and moderate to high disease activity by CDAI eligible for acceleration at Baseline that will have achieved low disease activity (LDA) by CDAI at 6 months in subjects treated in a T2T intervention group compared with a control group treated with usual care (UC), and to baseline disease activity.
4. To compare performance of derived outcome metrics between the T2T intervention and usual care at 6 and 12 months, including:

   1. DAS28 ESR
   2. Patient Reported Outcomes- RAPID 3
5. To determine the frequency of ineligibility for treatment acceleration due to risks, comorbidities, concomitant medication or clinician judgment in potential T2T study enrollees.
6. To compare rates of drug toxicities between the T2T and UC groups over 12 months.
7. To compare rates of Targeted Adverse Events (TAEs) between the T2T intervention and UC arms.

Exploratory Objectives To determine the rates and reasons for non-acceleration of subjects with qualifying CDAIs, enrolled in the T2T and UC arms.

Subjects with moderate to severe Rheumatoid Arthritis disease activity (defined as CDAI score >10) will be enrolled in the trial at participating sites. Sites will be randomized to either the Treat to Target or Usual Care arms. Visits will include a Baseline, Month 3, 6,9, and 12 visit for all subjects. In addition, subjects enrolled at sites participating in the Treat to Target Arm that have not achieved low disease activity (CDAI ≤10) will be expected to return for Monthly Assessment visits. Treatment acceleration will be expected to occur as frequently as monthly and at least every 3 months in these subjects, unless contraindicated.

Treatment acceleration for the purposes of this trial include the following options: Initiation or Change in prescribed treatment or dosage of "traditional" or "biologic" Disease Modifying Anti Rheumatic Drugs (DMARDs) or a change in the route of Methotrexate administration (from oral to subcutaneous)

Upon enrollment, physicians and subjects complete Enrollment Questionnaires, including a 28 joint assessment.

Targeted Adverse Event Reporting Qualifying adverse events which occur during participation in the study and are reported on the Targeted Adverse Event (TAE) Questionnaires. TAE Questionnaires are completed and submitted when a flagged event on a Physician Follow-up Questionnaire has been selected. Submission of de-identified source documents (i.e. hospital records, laboratory results, etc.) in support of the reported TAE is required in order to be valid, unless otherwise determined by the CORRONA Organization. The TAE should be simultaneously reported on both the TAE Questionnaire and on the CORRONA Data Collection Program Physician Follow-up Questionnaire visit date that most closely follows the event (unless the TAE occurs on the date of the Follow-up Visit).

In addition, sites will be encouraged to forward CORRONA, Inc.de-identified reports on qualifying Serious Adverse Events within 24 hrs of learning of them using the CORRONA SAE report form.

Data submitted for inclusion in the Database does not include the names, addresses, telephone numbers, email addresses, or social security numbers of subjects. Data from Questionnaires are tracked in the CORRONA Database by a unique CORRONA identifier assigned at the physician's office. A link is maintained at the physician's office between patient-identifying information (e.g., name, address, telephone number) and the unique CORRONA identifier. The physician's office does not share information with CORRONA that is needed to match subject names with these unique CORRONA identifiers.

Site Enrollment: Selected rheumatologists are invited to participate as investigators in the Treat to Target study.Not all rheumatologists who are involved in the CORRONA Data Collection Program will be involved in this study. Physicians are selected carefully to identify sites that have appropriate qualifications and infrastructure to support the trial and comply with applicable regulations and Good Clinical Practices to protect the rights of human subjects. All potential sites are screened for clinical research experience and GCP (Good Clinical Practice) training. Investigators must obtain Institutional Review Board (IRB) approval. Private physician offices and those not affiliated with an academic institution may submit to New England IRB (NEIRB). Sites at academic centers submit to their local institutional IRBs using approved templates and guidelines for submission, or to the NEIRB if this is approved by their institutional IRB.

Subject Informed Consent Informed consent will be obtained by the investigator and/or designee(s). Informed consent is obtained in the office setting, and in accordance with FDA regulations and guidelines prior to commencement of any study-specific related activities. Patient participation is voluntary, and participants may withdraw their consent at any time.

The CORRONA Organization conducts systematic reviews of submitted records. Additionally, all sites participating in the Treat to Target trial are expected to have at least one on-site monitoring visit during the course of the trial. This frequency may be adjusted, as needed, to address data quality issues.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the study will be both male and female adult (at least 18 years of age) patients who have a documented diagnosis of RA, are enrolled or willing to be enrolled in the CORRONA registry for the duration of the trial, have signed appropriate informed consent documents, are willing to participate in the trial, are medically appropriate for participation in the opinion of the investigator, and have moderate to severe RA disease activity as defined by CDAI >10.

Exclusion Criteria:

1. Patients under the age of 18
2. Women who are pregnant, breastfeeding or planning to become pregnant during the study period.
3. Patients with chronic or acute pain condition(s) other than active RA which, in the opinion of the investigator, is likely to confound or interfere with assessments of RA disease activity.
4. Functional class IV as defined by the ACR classification of functional status
5. Patients receiving a daily dose of prednisone of >10 mg within the 4 weeks prior to enrollment.
6. History of positive tuberculin skin test or equivalents that have not received documented treatment for latent tuberculosis (TB).
7. Patients with a significant, uncontrolled concomitant illness such as, but not limited to cardiovascular, renal, neurological, endocrinological, gastrointestinal, hepatic, metabolic, pulmonary or lymphatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Disease Activity, probability of treatment acceleration conditional on disease activity. | 1 year
  CDAI Score, rates of acceleration, frequency of visits, time to next visit conditional on disease activity, and probability of acceleration conditional on disease activity.

SECONDARY OUTCOMES:
Disease activity scores, reasons for ineligibility for treatment acceleration, frequency of toxicity, frequency of TAEs. | 1 year
  CDAI scores, DAS 28, RAPID 3, reasons/frequency of ineligibility for treatment acceleration, frequency of suspected (RA) drug-related toxicity, frequency of TAEs

CONTACTS AND LOCATIONS:
Overall Officials: Joel Kremer, MD, Principal Investigator — CORRONA, Inc.
Locations (1):
- The Center for Rheumatology, Albany, New York, United States

REFERENCES:
- [Derived] Harrold LR, Reed GW, Harrington JT, Barr CJ, Saunders KC, Gibofsky A, Greenberg JD, John A, Devenport J, Kremer JM. The rheumatoid arthritis treat-to-target trial: a cluster randomized trial within the Corrona rheumatology network. BMC Musculoskelet Disord. 2014 Nov 21;15:389. doi: 10.1186/1471-2474-15-389. PMID 25416400